CLINICAL TRIAL: NCT03183258
Title: Vascularised Sentinel Skin Flaps to Detect Rejection in Pancreas Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/SW/0333
Record Dates: First submitted 2017-06-05; First posted 2017-06-12 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Pancreas Transplant Rejection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel Skin Flap (Experimental)
  Interventions: Other: Sentinel skin flap

INTERVENTIONS:
Other: Sentinel skin flap — Donor-derived vascularised composite allograft (sentinel skin flap)

SUMMARY:
This pilot study aims to validate the use of vascularised donor-derived sentinel skin flaps for diagnosing rejection in pancreas transplantation. The aim of the study is to investigate the use of sentinel skin flaps in clinical practice and assess whether rejection occurs concordantly or discordantly between the skin flap and the transplanted abdominal organs. If successful, sentinel skin may allow improved immune surveillance and thereby facilitate earlier treatment of rejection with subsequent improvements in allograft survival and patient morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a pancreas transplant (SPK or PTA)
* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above

Exclusion Criteria:

* Patient does not have a patent ulna artery in either forearm
* Recipient of an enterically drained PTA
* Patient has received any investigational medical drug within 30 days of transplantation
* Patient is not willing to return to Oxford for all clinical follow-up for 12 months
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the trial, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05-19 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Concordant allograft rejection | 12 months
  If there is any clinical suspicion of rejection then both the sentinel skin flap and visceral allograft will be biopsied. Concordant rejection will be recorded where rejection is confirmed in both the sentinel skin flap and the visceral allograft.

SECONDARY OUTCOMES:
Discordant rejection of the sentinel skin | 12 months
  If there is any clinical suspicion of rejection then both the sentinel skin flap and visceral allograft will be biopsied. Discordant rejection will be recorded where there is rejection of the sentinel skin without rejection of the visceral allograft.
Discordant rejection of the visceral allograft | 12 months
  If there is any clinical suspicion of rejection then both the sentinel skin flap and visceral allograft will be biopsied. Discordant rejection will be recorded where there is rejection of the visceral allograft without rejection of the sentinel skin.
Donor specific antibodies | 12 months
  Development of de novo donor specific antibodies
Immunosuppression | 12 months
  Total dose immunosuppression
Graft survival | 12 months
  Pancreas allograft survival

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Friend, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom